CLINICAL TRIAL: NCT03464357
Title: Modification of Cortical Activation After Luminous Stimulation in Functional Magnetic Resonance Imaging (MRI) in Patients With Photophobia Related to Moderate to Acute Dry Eye Syndrome.
Brief Title: Functional MRI Study of Cortical Modifications to Light Stimulation in Patients With Photophobia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/17/0275; 2017-A02601-52 (Other: ID-RCB)
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Dry Eye Syndrome; Photophobia
Keywords: functional MRI
MeSH Terms: conditions — Dry Eye Syndromes; Photophobia

STUDY DESIGN:
Intervention Model Description: The study will compare the extent of neuronal activation at the visual cerebral cortex between a group with photophobia related to dry eye syndrome and a group of asymptomatic patients (without dry eye and no photophobia) with an MRIf.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symptomatic patients with dry eye (Active Comparator): 8 symptomatic patients with dry eye (mild to severe) assessed using a validated questionnaire (OSDI score, Appendix 1) associated with a disabling photophobia (need to wear sunglasses permanently outside, restriction of the outputs in case of significant brightness, restriction of the use of the screens because of the visual embarrassment ...). The fMRI will be carried out following the inclusion visit after all the necessary checks
  Interventions: Radiation: fMRI
- Asymptomatic patient (Active Comparator): 8 asymptomatic patients presenting neither photophobia (even minimal) or dry eye.
  The fMRI will be carried out following the inclusion visit after all the necessary checks
  Interventions: Radiation: fMRI

INTERVENTIONS:
Radiation: fMRI — The BOLD (Blood-Oxygen-Level Dependent) signal obtained by fMRI reflects the rate of oxygenation of the blood in the brain. However, the hemodynamic response that corresponds to an inflow of oxygenated blood increases in regions that consume energy. Thus, it is possible, by the study of the BOLD signal, to know with a great precision the regions of the brain specially active during a given task.
  The recorded signals reflect a neuronal activation. For each eye, recordings with and without flash visual stimulation are performed alternately.

SUMMARY:
Photophobia is a common and disabling symptom in patient with dry eye syndrome. The aim of this study is tried to better understand this complain analyzing brain activation during a luminous stimulation to highlight modification of cortical activation.

DETAILED DESCRIPTION:
Dry eye syndrome is a frequent and underestimated disease whose incidence tends to increase because of the population ageing and behaviors modification (time spent using screens increased, wearing of contact lenses…). Photophobia deteriorates the quality of life in patients with dry eye syndrome decreasing outdoor activities. This symptom is not understood and does not seem to be linked with dry eye syndrome severity. The study will compare cortical activation after luminous stimulation of 16 patients eyes (8 patients with dry eye syndrome and photophobia vs 8 asymptomatic patients) using functional MRI (fMRI).

The primary study endpoint was the extent of magnetic signals in visual cortex after luminous stimulation. Secondary endpoints were the spatial activation extent in the 3 areas of the visual cortex (Brodmann areas 17,18,19).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic subjects : presence of bilateral photophobia with an impact on daily activities (driving, outdoor activities, screens use, socio-professional activities…) in a context of patent dry eye syndrome
* Asymptomatic subjects : no dry eye syndrome and no photophobia
* Patients able to understand medical information and sign consent.

Exclusion Criteria:

* Ophthalmological pathologies of cornea, iris, optic nerve or retina
* MRI contraindications (metallic prosthesis, pacemaker, claustrophobia)
* Neurological pathology which may affect MRI results
* Subjects under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2018-03-13 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
The spatial extent of activation of the visual cortex | One day
  Measurement of voxel activation is validated and standardized (SPM8 software (Wellcome Department of Cognitive Neurology, London, UK) . In order to be able to determine the anatomical location of the voxels, a registration of the images on the standard image MNI152 (Montreal National Institute) provided by the Montreal Neurological Institute for which the spatial location of all the areas is known will be realized. It will thus be obtained, the number of activated voxels per visual area (Brodmann 17, 18, 19) for each hemisphere (contralateral and ipsilateral) of a subject with or without complaint.

CONTACTS AND LOCATIONS:
Overall Officials: François Malecaze, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No